CLINICAL TRIAL: NCT04914468
Title: Hamburg Transcatheter Mitral Valve Replacement Registry
Acronym: HERMES
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: HERMES
Record Dates: First submitted 2021-06-02; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Mitral Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Standardized methods for sample collection, processing, and storage, as well as appropriate storage facilities, are established and managed in accordance with the highest scientific and ethical standards. To ensure uniformity, quality, and reproducibility for the collection, processing, and storage of biomaterial, standard operating procedures (SOPs) are implemented.
  The following biomaterial will be sampled for additional biobanking within study visits:
  * Blood (whole blood, serum, plasma (EDTA, citrated,), DNA, RNA, washed erythrocytes
  * Urine
  * Tissue/ cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- TMVR: Patients undergoing Transcatheter Mitral Valce Replacement (TMVR)
- TEER: Patients undergoing mitral Transcatheter Edge-to-Edge Repair (TEER) after screening for TMVR
- Surgery: Patients undergoing mitral valve surgery (repair or replacement) after screening for TMVR
- Medical therapy: Patients undergoing medical therapy after screening for TMVR

SUMMARY:
The Hamburg TranscathEteR Mitral Valve REplacement RegiStry (HERMES) is a prospective clinical cohort registry aiming to gather follow-up information on short- and long-term outcome of patients with mitral valve disease that undergo transcatheter mitral valve replacement (TMVR) screening. In particular, long-term durability and function of implanted bioprosteses is of utmost interest for both patients and clinicians. Moreover, this study aimes to investigate and compare the different treatment strategies patients undergo after successful or unsuccessful screening for TMVR.

DETAILED DESCRIPTION:
Mitral valve regurgitation (MR) emerges as the most frequent valvular heart disease in developed coun-tries with prevalence increasing with age. Mitral valve repair is the gold standard therapeutic strategy in primary MR and is recommended in patients with secondary MR who are in need of revascularization. However, in patients with secondary MR mitral valve repair is associated with a higher rate of MR recurrence compared to mitral valve replacement. Nevertheless, elderly patients often are at high or prohibitive surgical risk and up to one half of all patients with severe MR are not referred to surgery. Transcatheter edge-to-edge mitral valve repair (TEER) constitutes a feasible and effective alternative, but eligibility for TEER is limited in some cases due to suboptimal anatomy or risk of mitral stenosis. Moreover, MR reduction is less predictable and, again, MR may reoccur. Transcatheter mitral valve replacement (TMVR) represents a complementary therapeutic approach for patients with severe MR. This novel therapy promises to reduce MR as durable as surgical valve replacement while reducing the procedural risk with an interventional approach.

The Hamburg TranscathEteR Mitral Valve REplacement RegiStry (HERMES) is a prospective clinical cohort registry aiming to gather follow-up information on short- and long-term outcome of patients with significant mitral valve disease, at high surgical risk with suboptimal anatomy for TEER, who undergo TMVR screening. In particular, long-term durability and function of implanted bioprosteses will be investigated. Additionally, this study aimes to investigate and compare the different treatment strategies patients undergo after successful or unsuccessful screening for TMVR (i.e., TMVR, TEER, surgery and medical therapy).

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent in accordance with Good Epidemiological Practice and local legislation.
* Individuals over the age of 18 years.
* Patients with clinically relevant mitral valve disease, who undergo screening for TMVR.

Exclusion Criteria:

* Insufficient knowledge of the German language, to understand study documents and interview without translation
* Physical or psychological incapability to cooperate in the investigation

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with clinically significant mitral valve regurgitation that undergo screening for Transcatheter Mitral Valve Replacement (TMVR) at University Heart and Vascular Center Hamburg shall be included. This includes inpatients and outpatients of the University Heart and Vascular Center Hamburg and may be extended to patients from other national or foreign centers. Inclusion into the study will take place after written informed consent is obtained. Patients included in interventional device studies (e.g., early feasibility TMVR studies, post-market TMVR studies etc.) may also be included in HERMES.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 6-60 months
  Incidence of death from any cause.
Cardiovascular mortality | 6-60 months
  Incidence of cardiovascular death, defined as death attributable to myocardial ischemia and infarction, heart failure, cardiac arrest because of other or unknown cause, or cerebrovascular accident.
Rehospitalization for congestive heart failure | 6-60 months
  Incidence of new-onset or worsening signs and symptoms of heart failure that required urgent therapy and resulted in hospitalization, e.g. as assessed by patient interviews.
Unplanned mitral valve intervention | 6-60 months
  Incidence of unplanned surgical or transcatheter re-intervention, heart transplantation or assist device implantation, e.g. as assessed by patient interviews.
Mitral regurgitation (MR) severity | 6-60 months
  Mitral regurgitation (MR) severity measured by transthoracic and/or transesophageal echocardiography. Assessment of MR severity according to current recommendations for valvular heart disease.

SECONDARY OUTCOMES:
Change in 6-minute-walking-test (6MWT) distance | 6-60 months
  6MWT will be performed by all participants at baseline and at follow-up visits.
Change in quality of life | 6-60 months
  Quality of life will be assessed by a standardized questionnaire [Kansas City Cardiomyopathy Questionnaire [KCCQ]) in all participants at baseline and at follow-up visits (or by phone interviews).
  The score is represented on a 0-to-100-point scale, where lower scores represent more severe symptoms and/or limitations and a score of 100 indicates no symptoms, no limitations, and excellent quality of life.
Change in New York Heart Association (NYHA) functional class | 6-60 months
  New York Heart Association [NYHA] functional class (I-IV) will be assessed in all participants at baseline and at follow-up visits (or by phone interviews).
  NYHA Class I: No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  NYHA Class II: Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  NYHA Class III: Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m). Comfortable only at rest.
  NYHA Class IV: Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Ludwig, MD, Principal Investigator — University Heart and Vascular Center Hamburg; Edith Lubos, MD, Principal Investigator — University Heart and Vascular Center Hamburg
Locations (1):
- University Heart and Vascular Center Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No